CLINICAL TRIAL: NCT05839951
Title: (STAR-T) Sequential TreAtment With Regorafenib and Trifluridine/Tipiracil (TAS-102, With or Without Bevacizumab) in Refractory Metastatic Colorectal Cancer: Real-world Outcomes in Community Clinical Practice in the USA
Brief Title: An Observational Study Called STAR-T to Learn More About the Sequential Treatment With Regorafenib and TAS-102 in Adults With Metastatic Colorectal Cancer Under Real World Conditions
Acronym: STAR-T
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22386
Record Dates: First submitted 2023-04-21; First posted 2023-05-03 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Colorectal Cancer (mCRC)
Keywords: Colon rectal cancer; Chemotherapy; Targeted medicine; Regorafenib; TAS-102
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms | interventions — regorafenib; trifluridine tipiracil drug combination; Trifluridine; tipiracil; Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort R-T: Patients with mCRC who started with regorafenib first, followed by TAS+/-Bev (Bevacizumab) without other therapies in between.
  Interventions: Drug: Regorafenib (BAY73-4506, Stivarga®); Drug: Bevacizumab
- Cohort T-R: Patients with mCRC who started with TAS+/-Bev first, followed by regorafenib, without other therapies in between.
  Interventions: Drug: TAS-102 (trifluridine and tipiracil, Lonsurf®); Drug: Bevacizumab
- Cohort TAS+BEV: Patients with mCRC who received combo use of TAS+BEV.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Regorafenib (BAY73-4506, Stivarga®) — Oral multitargeted kinase inhibitor
  Groups: Cohort R-T
Drug: TAS-102 (trifluridine and tipiracil, Lonsurf®) — Oral cytotoxic chemotherapy
  Groups: Cohort T-R
Drug: Bevacizumab — VEGFR inhibitor

SUMMARY:
This is an observational study using data that has been collected from participants who received their usual treatments.

Metastatic colorectal cancer (mCRC) is a cancer of the colon (large bowel) or the rectum (lowest part of the bowel just before the anus) that has spread to other parts of the body.

Regorafenib is an anti-cancer drug that blocks several proteins, called enzymes, which are involved in the growth of cancer. The combination of anti-cancer drugs trifluridine and tipiracil is called TAS-102. It prevents cancer cells from growing and multiplying.

Both regorafenib and TAS-102 are approved treatments for metastatic colorectal cancer and are available for doctors to prescribe to people with mCRC after previous lines of treatment have been unsuccessful.

Regorafenib and TAS-102 work in different ways and impact people differently. People might receive one of these drugs first and followed by the other. The best sequence for taking these drugs is still unclear.

Researchers have also found that TAS-102, when taken with another anti-cancer drug called bevacizumab, helps people live longer than when taken alone.

To better understand the impact of the sequence of taking regorafenib and TAS-102 (with or without bevacizumab), more knowledge is needed about how these work together in people with mCRC in real world settings.

The main purpose of this study is to learn more about the characteristics and impact of treatment in people with mCRC who received regorafenib and TAS-102 (with or without bevacizumab) one after the other. This information will be grouped based on their treatment sequence and age group (less or more than 65 years old).

In addition, the researchers want to learn about :

* how long participants were treated with regorafenib and TAS-102 taken one after the other in a sequential order,
* any treatment for mCRC that the participants received after the sequential treatment,
* any treatment received for a condition in which the bone marrow cannot make up enough blood cells (a common side effect of cancer treatment), during the sequential treatment,
* if and how often white blood cells that fight infection decreased during the sequential treatment,
* the number of hospital or testing facility visits that participants had during the sequential treatment, and
* how long did participants live (also called overall survival).

The participants in this study had already received regorafenib and TS-102 (with or without bevacizumab) as part of their regular care from their doctors.

The data will come from the participants' information stored in an electronic health records database called Flatiron mCRC EDM. Data collected will be from January 2015 to December 2022.

Researchers will only look at the health information from adults in the United States of America.

In this study, only available data from routine care is collected. No visits or tests will be required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who had diagnosis of mCRC (≥18 years old at diagnosis of mCRC)
* Received sequential treatment of regorafenib and TAS-102 (either mono or with bevacizumab) after mCRC diagnosis, with at least one documented clinical visit on or after treatment; OR
* Patients with mCRC who received combo use of TAS+BEV, with at least one documented clinical visit on or after treatment

Exclusion Criteria:

* Patients who had a diagnosis of gastrointestinal stromal tumors (GIST) or hepatocellular carcinoma (HCC) or other primary cancers in the baseline period (i.e., 6 months prior to index date) except non-melanoma skin cancers
* Patients involved in clinical trials during the study period (as indicated by the masked therapies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mCRC who received sequential treatment of Regorafenib and TAS-102 (with or without Bev), and patients with mCRC who received combo use of TAS+BEV from Jan 2015 to Sep 2022 (or 3 months prior to the latest data cut) from Flatiron CRC EDM data (v Dec 2022 or the latest version)
Sampling Method: Non-Probability Sample
Enrollment: 818 (Actual)
Dates: Start 2023-04-24 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Cohort R-T or Cohort T-R: Descriptive analysis of demographic | Retrospective analysis period is from Jan 2015 to Sep 2022 (or 3 months prior to the latest data cutoff date)
  Demographic includes age, gender, race and ethnicity, insurance.
Cohort R-T or Cohort T-R: Descriptive analysis of clinical characteristics | Retrospective analysis period is from Jan 2015 to Sep 2022 (or 3 months prior to the latest data cutoff date)
  Clinical characteristics includes number and type of prior therapies patient received for mCRC, stage at initial diagnosis, performance status, histology, time since metastatic diagnosis, Line of Treatment (LOT) of index treatment
Cohort R-T or Cohort T-R: Descriptive analysis of biomarker Kirsten rat sarcoma 2 viral oncogene homolog (KRAS) | Retrospective analysis period is from Jan 2015 to Sep 2022 (or 3 months prior to the latest data cutoff date)
  Biomarker B-Raf Proto-Oncogene (BRAF) and Mismatch Repair / Microsatellite instability (MMR/MSI) will be explored depending on data availability.

SECONDARY OUTCOMES:
Cohort R-T or Cohort T-R: Duration of sequential treatment | Retrospective analysis period is from Jan 2015 to Sep 2022 (or 3 months prior to the latest data cutoff date)
Cohort R-T or Cohort T-R: Proportion of patients receiving subsequent therapies | Retrospective analysis period is from Jan 2015 to Sep 2022 (or 3 months prior to the latest data cutoff date)
Cohort R-T or Cohort T-R: Type of subsequent therapies | Retrospective analysis period is from Jan 2015 to Sep 2022 (or 3 months prior to the latest data cutoff date)
Cohort R-T or Cohort T-R: Frequency of myelosuppression related medical interventions during sequential treatment | Retrospective analysis period is from Jan 2015 to Sep 2022 (or 3 months prior to the latest data cutoff date)
  Myelosuppression related medical interventions [e.g., use of Granulocyte colony stimulating factors (G-CSF)]
Cohort R-T or Cohort T-R: Frequency and incidence rate of neutropenia during sequential treatment | Retrospective analysis period is from Jan 2015 to Sep 2022 (or 3 months prior to the latest data cutoff date)
Cohort R-T or Cohort T-R: Number of patients with health care resource utilizations during sequential treatment | Retrospective analysis period is from Jan 2015 to Sep 2022 (or 3 months prior to the latest data cutoff date)
  Health care resource utilizations includes office/hospital visit and lab visit.
Cohort R-T or Cohort T-R: Overall survival of patients with Regorafenib followed by TAS-102 and vice versa in 3rd line treatment and 4th line treatment | Retrospective analysis period is from Jan 2015 to Sep 2022 (or 3 months prior to the latest data cutoff date)

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Whippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.